CLINICAL TRIAL: NCT01527513
Title: Effects of Eslicarbazepine Acetate (Esl, Bia 2-093) on Cognitive Function in Children With Partial Onset Seizures: an add-on, Double-blind, Randomised, Placebo-controlled, Parallel Group, Multicentre Clinical Trial
Brief Title: Effects of Eslicarbazepine Acetate (Esl, Bia 2-093) on Cognitive Function in Children With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-2093-208
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Partial Epilepsy
Keywords: Partial Epilepsy; eslicarbazepine acetate; Children
MeSH Terms: conditions — Epilepsies, Partial | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eslicarbazepine acetate (BIA 2-093) (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate (BIA 2-093) — Eslicarbazepine acetate (ESL) tablets 200 mg and the matching placebo will be supplied. Treatments will be administered by oral route, once-daily, in the evening. The dose will be rounded to the nearest 100 mg unit. Half tablets may be used for dose adjustment if necessary.
  Other Names: Eslicarbazepine acetate
  Arms: Eslicarbazepine acetate (BIA 2-093)
Drug: Placebo — Treatments will be administered by oral route, once-daily, in the evening.
  Arms: Placebo

SUMMARY:
To evaluate the effects of eslicarbazepine acetate on cognition in comparison with placebo as adjunctive therapy in children aged 6 to 16 years old with refractory partial-onset seizures.

DETAILED DESCRIPTION:
This will be a 2-part multicentre study in approximately 117 patients. Part I of the study will consist of a 4-week prospective observational baseline period, a 12-week double-blind period (4-week up-titration and 8-week maintenance), and a tapering-off period.

After the screening visit (V1), patients will enter the baseline period. At the end of the baseline period (V2), eligible patients will be randomised in a ratio of 2:1 to receive double-blind treatment with Eslicarbazepine acetate or Placebo in addition to concomitant therapy with 1 or 2 Anti-Epileptic Drugs (AEDs). Concomitant AED therapy will be kept stable during the whole study.

Initial dose of the study treatment will be 10 mg/kg/day. After 2-weeks on 10 mg/kg/day, the dose will be up-titrated to 20 mg/kg/day (maximum 1200 mg/day). After 2 weeks on 20 mg/kg/day, dose will be up-titrated to 30 mg/kg/day (maximum 1200 mg/day) and patients will receive this dose for 8 weeks. If intolerable adverse events (AEs) occur, the patient can be down-titrated to the previous dose (only 1 down-titration step will be allowed) or discontinued. After the 8-week maintenance period, the study treatment will be tapered off in 10 mg/kg/day 2 week steps. However, if a patient experiences an increase in seizure frequency (e.g. more than 100% increase vs. baseline) during tapering-off, the patient can proceed directly to the open-label part of the study (Part II).

After completion of the last 2-week 10 mg/kg/day step, patients will have the option to enter a 1 year open-label treatment (Part II) with Eslicarbazepine acetate (up to 30 mg/kg/day, maximum 1200 mg/day), or will have a 4 week observational follow-up period.

ELIGIBILITY:
Inclusion Criteria:

At visit 1 (screening), patient must be/have:

* written informed consent by parent or legal guardian and, where applicable, the patient;
* age 6 to 16 years, inclusive;
* a documented diagnosis of epilepsy for at least 12 months prior to screening;
* at least 2 partial onset seizures during the 4 weeks prior to screening despite treatment with 1 to 2 AEDs in a stable dose regimen;
* an Intelligence Quotient (IQ) of at least 70;
* current treatment with 1 to 2 AEDs (except oxcarbazepine, benzodiazepines other than clobazam and vagus nerve stimulation (VNS));
* excepting epilepsy, patient is judged to be in general good health based on medical history, physical examination and clinical laboratory tests;
* in the opinion of the investigator, able to complete the Cognitive Drug Research (CDR) test battery;
* in case of a girl of childbearing potential, patient presents a serum B-human chorionic gonadotropin (B hCG) test consistent with a non gravid state and agrees to remain abstinent or use reliable contraception (if used, hormonal contraception must be combined with a barrier method) starting at screening and continuing until at least the post-study visit (PSV).

At visit 2 (randomisation), patient must be/have:

* at least 2 partial-onset seizures during the 4 week baseline period prior to randomisation (documented in a diary);
* in case of a girl of childbearing potential, patient presents a urine B-hCG test consistent with a non-gravid state;
* stable dose regimen of concomitant AEDs during the 4 week baseline period;
* diaries satisfactorily completed by the patient or his/her caregiver during the baseline period;
* satisfactory compliance with the study requirements during the baseline period.

Exclusion Criteria:

At visit 1 (screening), patients must not be/have:

* only simple partial seizures with no motor symptomatology;
* primarily generalised seizures;
* known rapidly progressive neurological disorders (progressive brain disease, epilepsy secondary to progressive cerebral lesion);
* occurrence of seizures too close to count accurately;
* history of status epilepticus or cluster seizures (i.e., 3 or more seizures within 30 minutes) within the 3 months prior to screening; seizures of non-epileptic origin;
* Lennox-Gastaut syndrome;
* West syndrome;
* major psychiatric disorders;
* seizures of psychogenic origin within the last 2 years;
* history of schizophrenia or suicide attempt;
* history of attention deficit disorder or other diseases adversely affecting cognitive abilities;
* currently treated with oxcarbazepine, benzodiazepines other than clobazam (on a routine or chronic basis) and/or VNS;
* known hypersensitivity to carboxamide derivatives (oxcarbazepine or carbamazepine);
* uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological or oncology disorder;
* second or third degree atrioventricular blockade;
* relevant clinical laboratory abnormalities;
* estimated creatinine clearance (CLCR) <60 mL/min;
* pregnancy or nursing;
* treatment with eslicarbazepine acetate in any previous study;
* participation in other drug clinical trial within the last 2 months;
* not ensured capability to perform the trial;
* any other condition or circumstance that, in the opinion of the investigator, may compromise the patient's ability to comply with the study protocol.

At visit 2 (randomisation), patients must not be / have:

• any condition or circumstance that, in the opinion of the investigator, may compromise the patient's ability to comply with the study protocol.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- Italy (11):
  - Ospedale Salesi, Ancona
  - Ospedale Pediatrico Giovanni XXII, Bari
  - Ospedale Maggiore "C.A. Pizzardi", Bologna
  - Istituto Scientifico G. Gaslini, Genova
  - Ospedale Carlo Poma, Mantova
  - Policlinico Martino, Messina
  - Ospedale Fatebenefratelli, Milan
  - Policlinico Seconda Università di Napoli, Napoli
  - Istituto Mondino, Pavia
  - Ospedale Bambin Gesu, Roma
  - Azienda Ospedaliera O.I.R.M.- Sant'Anna, Torino
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Kempenhaeghe, location Heeze, Heeze
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Gabinet Lekarski Neurologii Dzieciecej i Leczenia Padaczki, Kielce
  - Wielkopolskie Centrum Neurologii Dzieci i Mlodziezy, Poznan
  - AKADEMIA MEDYCZNA im. Karola Marcinkowskiego w Poznaniu Katedra I Klinika Neurologii Wieku Rozwojowego, Poznan
  - Instytut "Pomnik-Centrum Zdrowia Dziecka", Warsaw
- Russia (11):
  - State Medical Institution "Children Republic Clinical Hospital of Minzdrav of Republic Tatarstan", Kazan'
  - Moscow State Healthcare Institution Scientific and Practical centre of medical help to children, Moscow
  - State Institution "Moscow Regional Scientific and Research Clinical Institute named after M.F. Vladimirsky", Moscow
  - OOO City Neurological Center "Sibneuromed", Novosibirsk
  - Saint Petersburg Scientific and Research Psycho-Neurology Institute, Saint Petersburg
  - Saint-Petersburg State Pediatric Medical Academy of Ministry of Health and Social development of Russian Federation, Saint Petersburg
  - Saint-Petersburg State Pediatric Medical Academy of Ministry of Health and Social, Saint Petersburg
  - Institution Russian Academy of Science Institute of human brain RAN, Saint Petersburg
  - Saint-Petersburg Sate Healthcare Institution "Children City Hospital #1", Saint Petersburg
  - State Healthcare Institution "Samarskaya Regional Clinical Hosptital named after M.I.Kalinin", Samara
  - Yaroslavskay State Medical Academy of Roszdrav, Yaroslavl
- Ukraine (7):
  - Donetsk Region Child Clinical Centre of Neuroreabilitation, Donetsk
  - Regional psycho-neurological hospital #3, Ivano-Frankivsk
  - chair of neuropathology and pediatric neurology of Kharkov Medical Academy, Kharkiv
  - Danylo Galytskyy Lviv National Medical University, Lviv
  - Communal institution "Child City Hospital #3", Odesa
  - Vinnytsya National Medical University,Vinnytsya Regional Psychoneurological Hospital, Vinnitsa
  - Zaporizhya regional clinical children hospital, Zaporizhzhya

REFERENCES:
- [Derived] Mintz M, Pina-Garza JE, Wolf SM, McGoldrick PE, Jozwiak S, Grinnell T, Cantu D, Costa R, Moreira J, Li Y, Blum D. Safety and Tolerability of Adjunctive Eslicarbazepine Acetate in Pediatric Patients (Aged 4-17 Years) With Focal Seizures. J Child Neurol. 2020 Mar;35(4):265-273. doi: 10.1177/0883073819890997. Epub 2019 Dec 26. PMID 31878820

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Once-Daily (QD)
- Esl (BIA 2-093): Eslicarbazepine acetate (BIA 2-093): ESL 10-30 mg/kg/day QD (maximum 1200 mg/day).
Period: Double Blind Period (DB) - Part I
Arm/Group | Placebo | Esl (BIA 2-093)
Started | 40 | 83
Randomized | 40 | 83
Safety Population | 40 | 83
Entered Maintenance Period | 40 | 76
Completed the Double Blind (DB)- Part I | 37 | 75
Eligible for Open Label Period (OL) | 37 | 75
Efficacy PP Population | 37 | 67
Per-protocol (PP) Population | 36 | 66
Completed | 37 | 75
Not Completed | 3 | 8
Period: Eligible for 1-Year Open Label Period
Arm/Group | Placebo | Esl (BIA 2-093)
Started | 0 | 112 (Participants that were eligible to participate in for 1-Year Open Label Period - Part II)
Completed | 0 | 95
Not Completed | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Esl (BIA 2-093): Eslicarbazepine acetate (BIA 2-093): ESL 30 mg/kg/day QD (maximum 1200 mg/day).
- Placebo: Placebo QD
- Total: Total of all reporting groups
Arm/Group | Esl (BIA 2-093) | Placebo | Total
Number analyzed (Participants) | 83 | 40 | 123
Age, Customized [Number; unit: participants]
  6-11 Years | 36 | 18 | 54
  12-16 Years | 47 | 22 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 14 | 50
  Male | 47 | 26 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 83 | 39 | 122
  South American | 0 | 0 | 0
  African (Black) | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Power of Attention Score to the End of the Double Blind (DB) Period
Description: Power of Attention was defined as the sum of the reaction time measures from the attentional tasks (simple [dominant hand only] reaction time, choice reaction time and digit vigilance speed) in order to assess information processing speed and attention/psychomotor speed.Change from baseline to the end of the double-blind period in Power of Attention will be compared between the treatment groups using an ANCOVA. Non-inferiority of ESL vs Placebo will be assessed by comparing the 95% CI's upper bound of the difference of Least Squares Mean (LSmeans) between treatment groups (ESL-placebo) with 121 ms. If the upper bound is greater than 121 ms then the null hypothesis that the change from baseline in the Power of Attention score in ESL group is at least 121 ms inferior than the placebo group will be rejected. Single Values were calculated the average of post treatment visits (visits 5 and 7or EDV) minus average of baseline visits (visits 1 and 2)
Time Frame: Visit 1 (-4 weeks for training), Visit 2 (Day 1), Visit 5 (6 weeks), Visit 7 (12 weeks) or at early discontinuation visit (EDV)
Population: The primary analysis was based on the Cognitive Per-protocol (PP) population - all patients in the Modified Cognitive Intent-to-Treat (ITT) population who completed the 8-week maintenance period and were not Important Protocol Deviations (IPDs) with respect to the primary cognitive endpoint.
Measure: Mean (Standard Error); unit: Milli seconds (ms)
Arm/Group | Placebo | Esl (BIA 2-093)
Number analyzed (Participants) | 34 | 60
Milli seconds (ms) | 111.085 (76.4254) | 59.122 (52.0904)
Statistical Analysis 1: Comparison: Placebo vs Esl (BIA 2-093); Test type: Non-Inferiority or Equivalence — A 121ms non-inferiority margin was selected based on a previous study with Cognitive Drug Research (CDR) system comparing newly diagnosed patients to a healthy normative sample. Assuming a Standard Deviation (SD) of 202.3 for the Power of Attention score, a total of 102 patients in the PP population would provide 80% power to reject the null hypothesis that the mean increase from baseline Power of Attention was at least 121 ms smaller in the placebo group; p = 0.700, 95% CI lower bound vs non-inf margin; Mean Difference (Final Values) = 33.2001, 95% CI 2-sided [-137.593 to 203.993]

2. Secondary Outcome: Change From Baseline in Standardized Seizure Frequency - Part I
Time Frame: Baseline; Titration Period (4 Weeks: V2-V3-V4)
Population: Modified Efficacy ITT population - all randomized patients who received at least one dose of study treatment after randomization and had at least one post-baseline seizure frequency assessment.
Measure: Mean (Standard Deviation); unit: Seizures per week
Arm/Group | Placebo | Esl (BIA 2-093)
Number analyzed (Participants) | 40 | 83
Seizures per week | -9.13 (75.602) | -31.03 (87.963)
Statistical Analysis 1: Comparison: Placebo vs Esl (BIA 2-093); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.700, ANCOVA; 95% CI lower bound vs non-inf margin = 33.2001, 95% CI 2-sided [-137.593 to 203.993] — The predefined non-inferiority margin was -121ms

3. Secondary Outcome: Change From Baseline in Seizure Frequency During the One-year Open-Label (OL)
Description: Overall Change from Baseline in Seizure Frequency per week for the One-Year Open-Label Period
Time Frame: Weeks 1 to ≥ 41 weeks
Population: Modified Efficacy Intent-to-Treat (ITT) population- all randomized patients who received at least one dose of study treatment after randomization and had at least one post-baseline seizure frequency assessment.
Measure: Mean (Standard Error); unit: Seizure per week
Groups:
- Esl PART II: Eslicarbazepine acetate (ESL) 10-30 mg/kg/day QD (maximum 1200 mg/day).
Arm/Group | Esl PART II
Number analyzed (Participants) | 112
Seizure per week | -3.03 (31.370)

ADVERSE EVENTS:
Time Frame: throughout the study
Groups:
- Part I - ESL; Part II - ESL: Eslicarbazepine acetate (ESL) - 30 mg/kg/day QD maximum 1200 mg/day.
Arm/Group | Placebo | Part I - ESL | Part II - ESL
Serious Adverse Events (participants affected / at risk) | 2/40 | 3/83 | 8/112
Other Adverse Events (participants affected / at risk) | 21/40 | 35/83 | 45/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Part I - ESL (N=83) | Part II - ESL (N=112)
ACUTE BRONCHITIS (Infections and infestations) | 1 | 0 | 0
INCREASED SEIZURE FREQUENCY OF COMPLEX MOTOR PARTIAL SEIZURES (Nervous system disorders) | 1 | 0 | 0
FRACTURE OF NOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0
MITRALIC INSUFFICIENCY (Cardiac disorders) | 0 | 1 | 0
COMPLEX PARTIAL STATUS (Nervous system disorders) | 0 | 1 | 0
Hepatitis infectious mononucleosis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Part I - ESL (N=83) | Part II - ESL (N=112)
Headache (Nervous system disorders) | 6 | 8 | 6
Somnolence (Nervous system disorders) | 2 | 5 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5 | 4
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Diplopia (Eye disorders) | 0 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 3 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 3 | 6
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Pyrexia (General disorders) | 2 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Astigmatism (Eye disorders) | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 3
Ear infection (Infections and infestations) | 0 | 1 | 2
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 3
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1
Varicella (Infections and infestations) | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Electrocardiogram t wave abnormal (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0
Hemianopia (Nervous system disorders) | 0 | 1 | 0
Mental retardation (Nervous system disorders) | 1 | 2 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Apathy (Psychiatric disorders) | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 2
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Hepatitis infectious mononucleosis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 4 | 3
Rubella (Infections and infestations) | 0 | 0 | 1
Scarlet fever (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 4
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other